CLINICAL TRIAL: NCT04219449
Title: Thrombophilia Versus Platelet Dysfunction In Beta Thalassemia
Brief Title: Thrombophilia In Beta Thalassemia
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, IM Yousef, Principal Investigator, Assiut University
Other Study IDs: TPDBT
Record Dates: First submitted 2019-12-27; First posted 2020-01-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Beta-Thalassemia
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: Diagnosed beta-thalassemia patients at Assiut University Hospital.
  Interventions: Diagnostic Test: PT; Diagnostic Test: Protein C; Diagnostic Test: Platelet aggregation by ADP and arachidonic acid

INTERVENTIONS:
Diagnostic Test: PT — measuring PT drawn on citrated blood sample
Diagnostic Test: Protein C — measuring protein C drawn on citrated blood sample
Diagnostic Test: Platelet aggregation by ADP and arachidonic acid — measuring platelet aggregation drawn on citrated blood sample

SUMMARY:
β-thalassemia disease is one of the most common congenital hemolytic anemia commonly found in the malarial belt areas including the Mediterranean, the Middle East, Africa, Southeast Asian countries, and China.

DETAILED DESCRIPTION:
β-thalassemia represents a major public health problem in Egypt, it is estimated that there are 1000/1.5 million per year live births born with β-thalassemia. The average life expectancy of patients with β-thalassemia has improved over the last few years as compared to that of in the previous millennium. This has led to the discovery of new set of problems such as increased hypercoagulable state in β-thalassemia like micro infarcts in spleen and lung indicating an activated coagulation pathway. The, incidence of thromboembolism in patients with thalassemia disease is approximately 10 times higher than normal population, it accounts between 1.7 and 9.2%. On the other hand, a study conducted by Chaudhary and Ahmad, 2012 showed decreased aggregation in majority of β-thalassemia patients. Another study conducted by Ibrahim, 1999 had noticed few patients to have bleeding manifestations in the form of epistaxis. Mussumeci et al., 1987 noted that both thrombophilic and anti-thrombophilic proteins were reduced as a consequence of liver damage. The net clinical outcome depends on the fine balance between the prothrombotic and antithrombotic pathways.

ELIGIBILITY:
Inclusion Criteria:

1. All blood samples from thalassemia patients before blood transfusion.
2. In splenectomized patients taking Aspirin, the tests will be performed 7 days after discontinuation of the drug.

Exclusion Criteria:

1. Patients with other hemoglobinopathies other than beta-thalassemia.
2. Patients suffering from hepatic or cardiac dysfunctions of another aetiology.
3. Patients with history of familial thrombophilia or use of anticoagulant therapy.

Ages: 4 Years to 20 Years | Sex: All
Age Groups: Child, Adult
Study Population: Diagnosed beta-thalassemia patients attending Pediatric Hematology Outpatient Clinic at Assiut University Hospital.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-07 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Hypercoagulability versus platelet dysfunction | one year
  Predominance of hypercoagulability versus platelet dysfunction in beta-thalassemia patients

SECONDARY OUTCOMES:
Regular screening of thalassemia patients | one year
  Evaluation of the significance of implementing regular screening of thalassemia patients for any possible hemostatic changes.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Winichakoon P, Tantiworawit A, Rattanathammethee T, Hantrakool S, Chai-Adisaksopha C, Rattarittamrong E, Norasetthada L, Charoenkwan P. Prevalence and Risk Factors for Complications in Patients with Nontransfusion Dependent Alpha- and Beta-Thalassemia. Anemia. 2015;2015:793025. doi: 10.1155/2015/793025. Epub 2015 Nov 18. PMID 26664743
- [Background] Cappellini MD, Motta I, Musallam KM, Taher AT. Redefining thalassemia as a hypercoagulable state. Ann N Y Acad Sci. 2010 Aug;1202:231-6. doi: 10.1111/j.1749-6632.2010.05548.x. PMID 20712798